CLINICAL TRIAL: NCT05805527
Title: Evaluating the Validity and Acceptability of a Fully-automated Interview to Diagnose Insomnia Disorder: a Pilot Study
Status: Completed | Type: Observational
Sponsor: University of Bordeaux (Other)
Responsible Party: Principal Investigator, Pierre Philip, Professor, University of Bordeaux
Other Study IDs: 0000
Record Dates: First submitted 2023-03-27; First posted 2023-04-10 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Insomnia Disorder
Keywords: Insomnia Disorder; Mobile health; Diagnosis
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: mobile health application named KANOPEE — Volunteers will undergo two clinical interviews, an in person clinician-led interview and a fully-automated interview administered via mobile phone

SUMMARY:
Objective: to evaluate if a fully-automated diagnostic interview for insomnia disorder is suitable for clinical and research purposes (adequate sensitivity and specificity) and is acceptable to patients.

Study main outcomes:

1. Concurrent validity (sensitivity and specificity) compared to a gold standard. Gold standard: clinical diagnosis of a clinician using a validated structured clinical interview for the DSM 5 criteria of insomnia disorder
2. Acceptability of the fully-automated interview.

Participants:

Volunteers to undergo the clinical and the automated interview will be recruited through non-probability convenience sampling from patients attending the sleep clinic at Bordeaux University Hospital between May 2023 and July 2023.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Being able to communicate and read in French
* Previous use a mobile phone

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteer patients attending the sleep clinic at the Bordeaux University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Concurrent validity (sensitivity and specificity) | May-July 2023
  Calculated with a gold standard evaluation consisting of the clinical diagnosis of a clinician using a validated structured clinical interview for the DSM 5 criteria of insomnia disorder

SECONDARY OUTCOMES:
Acceptability of the fully-automated interview | May-July 2023
  It will be measured with the Acceptability E-Scale (AES), that comprises six items and provides a total score as well as two subscores regarding usability (i.e. the perceived ease of using the system) and satisfaction with the system. Items are answered on a five-point Likert-type scale ranging from 1: Very unsatisfied, to 5: Very satisfied. Therefore, higher scores connote better acceptability.
Perceptions of the virtual agent | May-July 2023
  It will be measured with the ECA-Trust Questionnaire (ETQ), that includes six items that are answered on a four-point Likert-type scale ranging from 0: Not at all, to 3: Totally agree. It provides a total score as well as subscores on two separate dimensions, named perceived credibility and perceived benevolence of the virtual agent conducting the digital interview. Higher scores connote more trust.

CONTACTS AND LOCATIONS:
Overall Officials: Maria M Sanchez Ortuno, PhD, Study Director — Universite de Bordeaux, France - Universidad de Murcia, Spain
Locations (1):
- University Hospital of Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Philip P, Dupuy L, Morin CM, de Sevin E, Bioulac S, Taillard J, Serre F, Auriacombe M, Micoulaud-Franchi JA. Smartphone-Based Virtual Agents to Help Individuals With Sleep Concerns During COVID-19 Confinement: Feasibility Study. J Med Internet Res. 2020 Dec 18;22(12):e24268. doi: 10.2196/24268. PMID 33264099
- [Background] Auriacombe M, Fournet L, Dupuy L, Micoulaud-Franchi JA, de Sevin E, Moriceau S, Baillet E, Alexandre JM, Serre F, Philip P. Effectiveness and Acceptance of a Smartphone-Based Virtual Agent Screening for Alcohol and Tobacco Problems and Associated Risk Factors During COVID-19 Pandemic in the General Population. Front Psychiatry. 2021 Jul 16;12:693687. doi: 10.3389/fpsyt.2021.693687. eCollection 2021. PMID 34335332
- [Background] Dupuy L, Morin CM, de Sevin E, Taillard J, Salles N, Bioulac S, Auriacombe M, Micoulaud-Franchi JA, Philip P. Smartphone-based virtual agents and insomnia management: A proof-of-concept study for new methods of autonomous screening and management of insomnia symptoms in the general population. J Sleep Res. 2022 Apr;31(2):e13489. doi: 10.1111/jsr.13489. Epub 2021 Sep 18. PMID 34535942
- [Background] Philip P, Dupuy L, Sagaspe P, de Sevin E, Auriacombe M, Taillard J, Micoulaud-Franchi JA, Morin CM. Efficacy of a Smartphone-Based Virtual Companion to Treat Insomniac Complaints in the General Population: Sleep Diary Monitoring Versus an Internet Autonomous Intervention. J Clin Med. 2022 Jul 28;11(15):4387. doi: 10.3390/jcm11154387. PMID 35956005